CLINICAL TRIAL: NCT03456895
Title: Assessing Environmental Factors in Healthcare Facilities in Order to Improve the Experience of Patients, Staff, and the Quality of Imaging Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cincinnati (Other)
Collaborators: Ohio Third Frontier (Other); Wright Center of Innovation in Biomedical Imaging (Unknown)
Responsible Party: Principal Investigator, Michael V Knopp MD PhD, Professor, University of Cincinnati
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2017H0266/RP0525
Record Dates: First submitted 2018-01-05; First posted 2018-03-07 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Healthcare Facility Environment - Imaging
MeSH Terms: interventions — Auditory Perception; Smell

STUDY DESIGN:
Intervention Model Description: Three populations are being investigated in this trial; a healthy volunteer population, a patient population, and a staff population. Each population has the potential to participate in survey tools and/or physical environmental experiences.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy volunteer population (Experimental): Healthy volunteer participants will have one of two options for participation:
  1. completion of an electronic survey tool to assess the perception and preference of environmental factors (virtual participation)
  2. completion of the above survey and participation in environmental experiences and providing feedback about their experience (physical participation)
  Interventions: Other: Light perception; Other: Sound perception; Other: Smell perception; Other: Vibration perception; Other: Voice activation
- Patient population (Experimental): Patient participants will complete a survey tool and either participate in specific environmental experience testing or may be exposed to an environmental experience during the imaging examination. The imaging exam will be assessed in regard to quality factors such as motion artifacts as an indicator of being relaxed during the examination.
  Interventions: Other: Light perception; Other: Sound perception; Other: Smell perception; Other: Vibration perception; Other: Voice activation
- Staff population (Experimental): Staff participants who work in imaging-related healthcare environments will complete survey tools regarding their perception and preference of environmental factors and/or will participate in environmental experiences and provide feedback.
  Interventions: Other: Light perception; Other: Sound perception; Other: Smell perception; Other: Vibration perception; Other: Voice activation

INTERVENTIONS:
Other: Light perception — We will be using Wi-Fi/IP programmable LED lighting systems that will replace conventional lighting systems and may be in canned lights, spot lights, light chains or table lights. These lighting systems can be fully controlled by web based applications on smart phones tablets and computer systems and can be combined with input systems such as switches, motion detection or voice activated. Differences in lighting perception will be explored by varying lighting color and brightness.
Other: Sound perception — We will be using Wi-Fi/Bluetooth addressable sound systems that will be linked with sound sources such as media players on smart devices or computer systems. Differences in sound perception will be explored by varying sound types (i.e. different music types, ambient noise, etc.).
Other: Smell perception — We will explore the use of consumer grade ventilation systems that can be equipped to distribute packaged scents. Differences in smell perception will be explored by varying the types of scents.
Other: Vibration perception — We will explore the use of chairs or blankets that enable subjects to perceive vibrations. An initial implementation will be the use of on relaxing/massage chair that enables the experience of vibration sensation in the back or leg area. We may use also potentially vibration blankets in the arm or neck area. Differences in vibration perception will be explored by varying the location, frequency, etc. of vibrations with the subject being placed in a chair on an imaging table/bed.
Other: Voice activation — We will explore the use and linkage of voice activation system such as Amazon Echo, Google home or similar devices. Some participants may be asked to use voice activations to verbally select and/or change the environmental settings according to their preferences. We are evaluating the feasibility of voice activation with the imaging environment.

SUMMARY:
The purpose of this study is to assess subjects' perceptions of environmental conditions and their preferences, and to expose subjects to varied environmental conditions as well as to assess their perception and feedback to these conditions. Another aim of this study is to explore potential patterns, factors of influence, and factors of reference in relation to the objectively assessed quality of the imagining examination and/or the perception of the patient. Finally, another aim of this study is to explore the feasibility of innovative biofeedback response capturing methodologies and technologies to guide the design of specific clinical investigations or trials.

DETAILED DESCRIPTION:
Tremendous technological advances have occurred in recent years that enable easily controlled lights, sound, temperature, airflow as well as sensatory experiences such as smell or vibrations. While in some fields, these technologies are readily used, their potential application within healthcare environments has not yet been studied. In this study, we want to investigate how environmental factors including light, sound, temperature, smell, and sensatory experiences such as vibration are being perceived by subjects to develop environmental strategies using those components to create a more relaxing, and comforting experience for patients prior, during and after an imaging examination and for staff working in such environments. This data that will also guide to encourage changes of patient staff facility interactions to further improve the healthcare experience and quality of imaging examinations. To get a complete set of data, we plan to include volunteer participants, patients scheduled for imaging examinations, and staff working in the healthcare environment. This study has up to three different components: A, filling out survey forms to learn more about the perception of experience factors B, participating in facility experiences that may expose subjects to different facility factors and will then assess responses using additional survey forms or electronic measurement and data capture devices and C, during an imaging study the environment experience may be altered and assessments will be done to determine how relaxed the subject remains during the imagining study and the degree of motion induced artifacts. Feedback data will be obtained through survey tools as well as available consumer grade wearable devices that can continuously capture physiological parameters such as heart rate, motion, body perspiration and muscle tension. Only participants in the patient, staff, or volunteer populations who are not receiving an MRI imaging examination will participate in utilizing the wearable devices, as the wearable devices are not compatible with the MRI system. Patients receiving a PET/CT examination will be able to utilize a wearable device. For patients scheduled for an imaging examination the findings and perception of environmental factors will be compared with the image quality of the imaging examination and the feedback responses.

ELIGIBILITY:
Inclusion Criteria:

Volunteer population:

- Male and female volunteers above the age of 18 who are able to give an informed consent or have a legal guardian able to give informed consent on their behalf

Staff population:

- Male and female staff at the Ohio State University above the age of 18 who are able to give informed consent

Patient population:

* Male and female patients greater than or equal to 18 years of age able to give informed consent or have a guardian able to give informed consent on their behalf
* Patients must have an imaging study such as an MRI, PET/CT, or CT scheduled to be performed at the Wright Center facility at Martha Morehouse

Exclusion Criteria:

* Unable to communicate in English
* Subjects that are incapable of giving informed consent or that do not have a legal guardian to give informed consent on their behalf.
* Prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mood, Physiological State - Heart Rate | Participants may complete physiological measurements through study completion, on average 1 year.
  Participants' mood will be assessed via measurements of participants' heart rate
Mood, Physiological State - Body Temperature | Participants may complete physiological measurements through study completion, on average 1 year.
  Participants' mood will be assessed via participants' body temperature
Mood, Self-Report | Participants may complete surveys through study completion, on average 1 year.
  Participants' mood will be assessed via self report in surveys
Environmental preference | Participants may complete surveys through study completion, on average 1 year.
  Participants will self-report their preferences for different light, sound, smell, and vibration sensations
Feasibility of the use of voice activation within the imaging environment | We will be observing the feasibility of voice activation through study completion, on average 1 year.
  We are observing how practical and beneficial it is to use voice activation technologies such as Amazon Echo, Google home or similar devices within the imaging environment. For instance, we will observe how user-friendly, time-consuming, etc. the use of voice activation technology is within an imaging setting for assessing participant preferences.

SECONDARY OUTCOMES:
Temperature | Temperature of the environment and of each participant may be monitored from the time the participant begins the environmental experience until the participant completes study procedures, up to roughly 1 hour
  We will use infrared detector camera technology to assess the skin temperature of subjects at different body regions and changes during the observational period. This will also be used to determine the temperature of the surroundings as well, for example, to determine the relative temperature of the chair and the imaging bed. Infrared cameras installed alongside the normal surveillance cameras to monitor patients during the imaging examination may also be used to monitor the temperature of the surroundings as well as the body to determine if that may be the reason for motion.
Motion | Motion of each participant may be monitored from the time the participant begins the environmental experience until the participant completes study procedures, up to roughly 1 hour
  We will use short wave radar to perform positional monitoring of subjects during the observational period. This short-wave radar will be used as a means to assess motion and detect subject movement in a room that we hope to correlate to their level of comfort and relaxation. Short wave radar is also technically able to detect very miniscule motion including blood flow and pulse rate, which would allow us to move away from wearable devices to remote sensing devices further hoping to increase patient comfort. No short wave radar devices will be used during the imaging examination.
Quality of imaging study | Image quality will be assessed after SOC images are collected from patient participants through study completion, on average 1 year.
  Patient participants who have given authorization for a blinded review of their imaging study will have their imaging study reviewed on a radiological image review workstation and assessed by an experienced reader of imaging studies in regard to the presence and severity of artifacts. Those findings will be recorded both in a structured and free text form using a survey tool. We anticipate that in this exploratory study observations will be made that will lead to the need to further detail and/or refine structured recording of the findings.

CONTACTS AND LOCATIONS:
Overall Officials: Michael V Knopp, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Knopp MU, Binzel K, Wright CL, Zhang J, Knopp MV. Enhancing Patient Experience With Internet Protocol Addressable Digital Light-Emitting Diode Lighting in Imaging Environments: A Phase I Study. J Med Internet Res. 2020 Jun 12;22(6):e11839. doi: 10.2196/11839. PMID 32530434

DOCUMENTS (1):
  • Study Protocol (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT03456895/Prot_000.pdf